CLINICAL TRIAL: NCT02826759
Title: Comparison of Serum Sphingolipidomic Analyses in Healthy, Pre-diabetic and Diabetic Subjects
Brief Title: Serum Sphingolipidomic Analyses in Healthy, Diabetic and Prediabetic Subjects
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: KYLLSL201312701; 13040470432 (Other Grant/Funding Number: Chinese Medical Association); 2013YK20 (Other Grant/Funding Number: The First Affiliated Hospital of Xi'an Jiaotong University)
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2; Prediabetic State
Keywords: sphingolipid; diabetes mellitus; biomarker; obesity; insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Diabetes Mellitus; Obesity; Insulin Resistance | interventions — insulin resistance factor (uremia)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples are used to test the concentration of sphingolipid metabolites ( ceramide, sphingosine, sphingosine-1-phosphate, sphinganine, sphinganine-1-phosphate) by mass spectrometry
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- serum sphingolipid metabolites in healthy subjects: Healthy subjects are classified according to BMI into three subgroups: healthy normal weight subjects, healthy overweight subjects and healthy subjects with obesity. Age and sex are matched among three subgroups. serum sphingolipid metabolites including sphingosine-1-phosphate will be compared.
- serum sphingolipid metabolites in diabetic subjects: Diagnosed diabetic patients are divided into three subgroups: diabetic patients with normal weight, overweight and obesity. age and sex are matched.
  Interventions: Other: diabetes
- serum sphingolipid metabolites in the progression of diabetes: serum sphingolipid metabolites are compared among three age-, sex- and body mass index-matched subgroups: healthy subjects, subjects with pre-diabetes, subjects with diabetes
  Interventions: Other: diabetes
- serum sphingolipid metabolites and HbA1c: diabetic subjects are divided by HbA1c level. the cut-offs are 7% and 9%. serum sphingolipid metabolites will be tested among diabetic patients with HbA1c <7%, 7%-9% and >9%
  Interventions: Other: diabetes
- serum sphingolipid metabolites in insulin-resistant subjects: comparison of serum sphingolipid metabolites in newly diagnosed insulin-resistant subjects and age-, sex- and BMI-matched healthy controls.
  Interventions: Other: diabetes

INTERVENTIONS:
Other: diabetes — the exposure of interests are obesity, diabetes and insulin-resistance
  Other Names: insulin-resistance
  Groups: serum sphingolipid metabolites and HbA1c; serum sphingolipid metabolites in diabetic subjects; serum sphingolipid metabolites in insulin-resistant subjects; serum sphingolipid metabolites in the progression of diabetes

SUMMARY:
This study is designed to compare the serum sphingolipidomic analyses in healthy, pre-diabetic and diabetic subjects. age, sex and BMI are matched among these three groups. As ceramide, sphingosine, sphingosine-1-phosphate and sphinganine are involved in inflammation, immunity and cancer, investigators proposed a hypothesis that sphingosine-1-phosphate and other sphingolipids may be associated with the progress of type 2 diabetes. sphingolipids may be a biomarker for diabetes.

DETAILED DESCRIPTION:
The first purpose of this study is to determine whether serum sphingolipid metabolites associate significantly with the weight among type 2 diabetes. 60 patients with diagnosed type 2 diabetes will be recruited. The serum concentrations of sphingolipid metabolites of 20 type 2 diabetic patients with obesity will be compared to age- and sex-matched series of 40 type 2 patients without obesity.

The second purpose of this study is to determine whether serum sphingolipid metabolites associate significantly with the process and severity of type 2 diabetes. The serum concentrations of sphingolipid metabolites of 20 subjects with type 2 diabetes will be compared to age-, sex- and BMI-matched series of healthy and pre-diabetic subjects. Investigators speculate that the serum concentration of sphingolipid metabolites are positively related with the progression of diabetes. In order to discover why serum sphingolipid metabolites correlates with the progression of diabetes, detailed information on HbA1c, duration of diabetes history and insulin resistance defined by homeostatic model assessment (HOMA-IR) will be analysed. These three parameters may affect the serum concentrations of sphingolipid metabolites.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of diabetes mellitus, type 2
* clinical diagnosis of prediabetic status
* older than 18 and younger than 90 years-old
* clinical diagnosis of insulin-resistance
* clinical diagnosis of newly onset of diabetes mellitus, type 2
* those who are willing to participate in the trial and sign the consent form

Exclusion Criteria:

* any cardiovascular disease (myocardial infarction, heart failure, cerebrovascular accident)
* missing information of BMI
* sever liver, kidney dysfunction
* sever pancreatitis or those who received pancreatectomy
* on medications of hormone, immunosuppressive therapy or drugs that may affect the bioactivity or concentration of sphingolipids (e.g. asprin )
* patients on pregnancy
* sever systematic diseases including carcinoma, mental disorder, sever anemia et al.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects undergoing oral glucose tolerance test and hospitalized type 2 diabetic patients in the Dpartment of Endocrinology in the First Affiliated Hospital of Xi'an Jiaotong Unversity are collected.
  healthy subjects undergoing routine physical exam in the department of medical examination center, First Affiliated Hospital of Xi'an Jiaotong Unversity are recruited
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
serum concentration of sphingosine-1-phosphate, micromol per liter | Nov, 2016

SECONDARY OUTCOMES:
serum concentration of sphingosine, micromol per liter | Nov, 2016
serum concentration of sphinganine-1-phosphate, micromol per liter | Nov, 2016
serum concentration of sphinganine, micromol per liter | Nov, 2016
serum concentration of ceramide, micromol per liter | Nov, 2016

CONTACTS AND LOCATIONS:
Overall Officials: Jing Sui, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Sui J, He M, Wang Y, Zhao X, He Y, Shi B. Sphingolipid metabolism in type 2 diabetes and associated cardiovascular complications. Exp Ther Med. 2019 Nov;18(5):3603-3614. doi: 10.3892/etm.2019.7981. Epub 2019 Sep 6. PMID 31602237